CLINICAL TRIAL: NCT07078760
Title: Lattice-tip Versus Irrigated-tip Catheter for Linear Ablation of the Cavotricuspid Isthmus. A Multicenter, Randomized Study. (The LINEAR Study)
Brief Title: Lattice-tip Versus Irrigated-tip Catheter for Linear Ablation of the Cavotricuspid Isthmus. A Multicenter, Randomized Study.
Acronym: LINEAR
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mitera Hospital (Other)
Responsible Party: Principal Investigator, Stylianos Tzeis, MD, PhD, FEHRA, Cardiologist - Electrophysiologist, Mitera Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 833α/ΔΣ
Record Dates: First submitted 2025-07-04; First posted 2025-07-22 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Catheter Ablation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CTI radiofrequency ablation with lattice-tip catheter (Active Comparator): Patients undergoing CTI catheter ablation using RF energy delivered by the lattice-tip, dual-energy catheter (Sphere-9, Medtronic).
  Interventions: Procedure: CTI radiofrequency ablation.
- CTI radiofrequency ablation performed with irrigated-tip catheter (Active Comparator): Patients undergoing CTI catheter ablation using RF energy delivered by the irrigated RF catheter (ThermoCool® SmartTouch™, Biosense Webster, USA).
  Interventions: Procedure: CTI radiofrequency ablation.

INTERVENTIONS:
Procedure: CTI radiofrequency ablation. — Cavotricuspid Isthmus ablation

SUMMARY:
The LINEAR study is designed to compare the procedural efficacy, efficiency and safety of linear radiofrequency ablation of the cavotricuspid istmus using either a standar irrigated-tip ablation catheter or lattice-tip ablation catheter .The primary focus of the acute procedural data analysis will be:

Procedural efficacy: This will be evaluated based on the rate of bidirectional CTI block persistence after 60 min waiting period documented by high resolution activation mapping. Furthermore, provocative test with intravenous adenosine infusion will be conducted to exclude dormant CTI conduction.

Procedural efficiency: This will be evaluated based on the number of RF lesions delivered, time to achieve bidirectional CTI block, and fluoroscopy exposure time.

Procedural safety: The incidence of procedural complications will be recorded.

DETAILED DESCRIPTION:
This is a prospective, multicenter, randomized controlled trial designed to compare the efficacy, efficiency and safety of CTI catheter ablation using two different catheter technologies: the lattice-tip, dual-energy catheter (Sphere-9, Medtronic) and the irrigated radiofrequency (RF) catheter (ThermoCool® SmartTouch™, Biosense Webster, USA). The primary focus of the acute procedural data analysis will be:

Procedural efficacy: This will be evaluated based on the rate of bidirectional CTI block persistence after 60 min waiting period documented by high resolution activation mapping. Furthermore, provocative test with intravenous adenosine infusion will be conducted to exclude dormant CTI conduction.

Procedural efficiency: This will be evaluated based on the number of RF lesions delivered, time to achieve bidirectional CTI block, and fluoroscopy exposure time.

Procedural safety: The incidence of procedural complications will be recorded.

Patient Population Based on previously published data, the proportion of patients with documented CTI bidirectional block at 60 minutes as assessed by high density electroanatomical mapping is estimated at 60% for the control group. Based on preliminary studies conducted by our group, we expected a respective percentage of bidirectional block of 85% in the intervention group. Hence, for a superiority design with two-sided α of 0.05, equal (1:1) allocation between groups and 80% power, 48 patients per group (96 in total) were estimated as the target sample size. As the outcome is assessed intraprocedurally, no dropouts are expected, and therefore no further adjustments were made to the sample size estimations.

Patients will be prospectively randomized in a 1:1 ratio to one of two treatment groups:

* Group A: Patients undergoing CTI catheter ablation using RF energy delivered by the lattice-tip, dual-energy catheter (Sphere-9, Medtronic).
* Group B: Patients undergoing CTI catheter ablation using RF energy delivered by the irrigated RF catheter (ThermoCool® SmartTouch™, Biosense Webster, USA).

Ablation Procedure All participants will receive anticoagulation therapy for a minimum of one month prior to the ablation procedure. All anti-arrhythmic drugs (AADs) will be discontinued at least five half-lives before the procedure. General anesthesia (GA) will be utilized in both groups.

A decapolar electrode catheter will be positioned in the coronary sinus (CS) before the commencement of ablation. In patients presenting with sinus rhythm, ablation will be performed during pacing from the proximal CS bipole at a cycle length of approximately 600 ms. For patients presenting with typical atrial flutter, pacing will be initiated following termination of the flutter.

CTI ablation will be performed using a point-by-point catheter technique, creating a contiguous line of lesions along the CTI, guided by fluoroscopy, electroanatomical mapping. The catheter will be gently dragged from the tricuspid valve annulus towards the inferior vena cava. Intracardiac echocardiography (ICE) will be utilized as an adjunct in cases where bidirectional block is not readily achieved, to further evaluate potential anatomical variations.

In Group A, only RF energy will be delivered using the dual-energy focal 9 mm lattice-tip catheter (Sphere-9; Medtronic) according to the recommended settings. Pulsed field ablation will not be employed in this group.

In Group B, the VISITAG module will be utilized to tag the location of each RF lesion application, with the following settings: stability range of 2-3 mm, stability duration of 3-5 s, force over time of 25%, and a tag size diameter of 3 mm. The power setting will be at 30 W with a target contact force of 10-30 g and a target Ablation Index value of 400. Saline irrigation will be administered at a rate of 30 mL/min, and the temperature limit will be set at 43 °C.

Primary Efficacy Endpoint The primary procedural endpoint for efficacy will be the achievement of bidirectional CTI block. After completion of the CTI line, bidirectional block will be confirmed through differential pacing maneuvers followed by activation mapping, performed using the Affera mapping system for Group A and the CARTO mapping system for Group B, respectively. Activation mapping will be repeated 60 minutes after the initial documentation of bidirectional block to assess for its persistence or the presence of spontaneous recovery of CTI conduction

Primary Safety Endpoint The incidence of procedural complications will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* patients above 18 years of age undergoing CTI ablation

Exclusion Criteria:

* Prior right atrium ablation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Estimated)
Dates: Start 2025-06-16 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The primary procedural endpoint for efficacy will be the achievement of bidirectional CTI block after 60 min waiting period documented by high resolution activation mapping . The primary safety endpoint will be the incidence of procedural complications. | 60 minutes
  The primary procedural endpoint for efficacy will be the achievement of bidirectional CTI block. After completion of the CTI line, bidirectional block will be confirmed through differential pacing maneuvers followed by activation mapping, performed using the Affera mapping system for Group A and the CARTO mapping system for Group B, respectively. Activation mapping will be repeated 60 minutes after the initial documentation of bidirectional block to assess for its persistence or the presence of spontaneous recovery of CTI conduction. In the absence of spontaneous recovery, a provocative test involving intravenous adenosine infusion will be conducted to evaluate for dormant CTI conduction. During the adenosine infusion and the resultant transient atrioventricular block or sinus pause, bidirectional block will be reassessed using differential pacing maneuvers with the mapping catheter positioned laterally to the ablation line.The incidence of procedural complications will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Stylianos Tzeis, MD, PhD, FEHRA, Principal Investigator — Mitera Hospital
Locations (1):
- Mitera General Hospital, Athens, Attikis, Greece

IPD SHARING:
Plan to Share IPD: Undecided